CLINICAL TRIAL: NCT03168204
Title: Study Protocol of the D-SCOPE Project With a Randomized Controlled Trial, Evaluating the Efficacy of a Detection and Prevention Program for Frail Community-dwelling Older Adults
Brief Title: Evaluating the Efficacy of a Detection and Prevention Program for Frail Community-dwelling Older Adults
Acronym: D-SCOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Hogeschool Gent (Unknown); Universiteit Antwerpen (Other); KU Leuven (Other); Maastricht University (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Principal Investigator, Liesbeth De Donder, Prof. Dr. Liesbeth De Donder, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D-SCOPE IWT 140027
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Older Adults
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Risk of being frail experimental group (Experimental)
  Interventions: Behavioral: Tailored care and support
- Risk of being frail control group (No Intervention)
- No/low risk of being frail (No Intervention)
- Risk of being frail care avoiders (No Intervention)

INTERVENTIONS:
Behavioral: Tailored care and support — Offering tailored care and support whereby the competences, strengths and resources of the older person are taken into account.The intervention will be an enhancement of usual care and will depend on the availability of the municipality, and could be formal (i.e., home care) or informal (e.g. activities of an older adult's association).
  Arms: Risk of being frail experimental group

SUMMARY:
The evaluation of a detection and prevention program which aims to create a continuum of care and support for frail community-dwelling older people (from early detection, over intervention, to follow-up). First, the program aims to develop methods to easily, accurately and timely detect and prevent a negative frailty-balance in older people. Second, the study aims to improve the quality and efficacy of care and support given to frail community-dwelling older people.

ELIGIBILITY:
Inclusion Criteria:

Sample 1: 150 older people per municipality (total: 3 municipalities) (inclusion criteria: at least one selection criterion)

* Gender: 75 men - 75 women
* Age: 25 older people aged between 60 and 70 years old - 125 older people older than 70 years
* Marital status: 50 older people with partner - 100 older people without partner
* Living situation: 100 older people who have not moved last 10 years - 50 older people who have moved last 10 years
* Migration background: 100 older people born in Belgium - 50 older people born elsewhere

Sample 2: 150 older people per municipality (total: 3 municipalities) (inclusion criteria: all selection criteria at once)

* 75 men, older than 70 years, living together/widowed/divorced/never married, moved last 10 years
* 75 women, older than 70 years, widowed/divorced/never married, moved last 10 years

Exclusion Criteria:

* Current institutionalization
* Current hospitalization

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 869 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline Quality of Life at 6 months | Assessed during baseline testing + 6 months after inclusion
  One question from the WHOQOL-BREF will be used to measure the quality of life of participants (1 item). Older participants will also be asked to rate their quality of life on a scale from 0 to 10.
Change from baseline Satisfaction with Life at 6 months | Assessed during baseline testing + 6 months after inclusion
  The Satisfaction with Life Scale will be administered to explore the life satisfaction of the participants (5 items)
Change from baseline sense of mastery at 6 months | Assessed during baseline testing + 6 months after inclusion
  To assess the sense of mastery of older people, the current mastery questionnaire will be used and one self-constructed item will be added which will assess mastery in relation to others. Older participants will also be asked to rate their mastery on a scale from 0 to 10.
Change from baseline Meaning in Life at 6 months | Assessed during baseline testing + 6 months after inclusion
  Meaning in life will be evaluated with 5 items from the Meaning in Life Questionnaire (MLQ). Older participants will also be asked to rate their meaning in life on a scale from 0 to 10.
Change from baseline Community Inclusion at 6 months | Assessed during baseline testing + 6 months after inclusion
  Community inclusion will be measured using 1 item from the Community Integration Measure (CIM). Older participants will also be asked to rate their community inclusion on a scale from 0 to 10.
Change from baseline aging well in place at 6 months | Assessed during baseline testing + 6 months after inclusion
  One self-constructed question (1 item) will assess if the older person lives at home in a qualitative manner

SECONDARY OUTCOMES:
Multidimensional frailty | Assessed during baseline testing + 6 months after inclusion
  The Comprehensive Frailty Assessment Instrument (CFAI) will be used to measure multidimensional frailty: physical, cognitive, psychological, social and environmental frailty
Physical phenotype of frailty | Assessed during baseline testing + 6 months after inclusion
  The Fried's phenotype of frailty will be used to assess the physical phenotype of frailty as well as the questionnaire of Op het Veld
Feeling frail | Assessed during baseline testing + 6 months after inclusion
  The subjective feeling of frailty will be assessed using 1 self-constructed question and will assess to what extent an older person feels frail
Resilience | Assessed during baseline testing + 6 months after inclusion
  Resilience will be measured using the Connor-Davidson Resilience Scale (CD-RISC2), which is an abbreviated 2-item version of the original scale
Coping | Assessed during baseline testing + 6 months after inclusion
  Coping will be measured using 12 items from the BRIEF cope. Two items from active coping, positive reframing, religion, use of emotional support and self-distraction and one item from acceptance and behavioral disengagement will be used
Help needed for activities in daily life | Assessed during baseline testing + 6 months after inclusion
  Older people will be asked if they need help with 8 activities of daily life, and to what extent the help they receive for these activities is sufficient. These questions are adapted from the questionnaire of the Belgian Ageing Studies (BAS)
Informal and formal care | Assessed during baseline testing + 6 months after inclusion
  Older people will be asked if they receive care from 6 informal and 14 formal caregivers and if they are satisfied with the help they receive from these caregivers. These questions are adapted from the BAS-questionnaire.
Medical care | Assessed during baseline testing + 6 months after inclusion
  The participants will be asked if they needed to go to the hospital, to a residential setting and a rehabilitation center over the past 6 months (day case/overnight stay). These questions are adapted from the Health Interview Survey. In addition, the participants will be asked when they visited the general practitioner for the last time over the last 6 months.
Leisure time | Assessed during baseline testing + 6 months after inclusion
  Leisure time will be measured by using an adapted question with 8 items derived from the BAS-questionnaire and will examine how often the participants perform the listed activities
Neighborhood | Assessed during baseline testing + 6 months after inclusion
  Different dimensions of neighborhood will be assessed. First, the social environment will be administered by using 3 items from the social cohesion dimension of the Neighbourhood Scale. Second, the physical environment will be explored by using 4 items from the BAS-questionnaire as well as from the Neighbourhood Environment Walkability Scale. Finally, low-key participation will be examined by using 2 items from the questionnaire of Oswald & Konopik.
Life-events | Assessed during baseline testing + 6 months after inclusion
  A shortened version of the Geriatric Adverse Life Events Scale (GALES) will be adapted to assess to occurrence of life-events (11 items)

CONTACTS AND LOCATIONS:
Overall Officials: Liesbeth De Donder, Prof. Dr., Principal Investigator — Vrije Universiteit Brussel
Locations (3):
- Belgium (3):
  - OCMW Gent, Ghent
  - OCMW Knokke-Heist, Knokke-Heist
  - OCMW Tienen, Tienen

REFERENCES:
- [Derived] Van der Elst M, Schoenmakers B, Dierckx E, De Donder L, De Roeck E, Duppen D, Fret B, Schols JMGA, Kempen GIJM, De Lepeleire J. A search for relevant contextual factors in intervention studies: a stepwise approach with online information. BMJ Open. 2022 Sep 9;12(9):e057048. doi: 10.1136/bmjopen-2021-057048. PMID 36691193
- [Derived] Dierckx E, Duppen D, Hoens S, Switsers L, Smetcoren AS, De Donder L, D-Scope. Effectiveness, satisfaction and meaningfulness of a 6-step detection and prevention program for frail community-dwelling older adults: a mixed-method evaluation. BMC Geriatr. 2022 Dec 14;22(1):966. doi: 10.1186/s12877-022-03504-7. PMID 36517745
- [Derived] Lambotte D, De Donder L, De Roeck EE, Hoeyberghs LJ, van der Vorst A, Duppen D, Van der Elst M, Fret B, Dury S, Smetcoren AS, Kardol MJM, Engelborghs S, De Deyn PP, De Witte N, Schols JMGA, Kempen GIJM, Zijlstra GAR, De Lepeleire J, Schoenmakers B, Verte D, Dierckx E. Randomized controlled trial to evaluate a prevention program for frail community-dwelling older adults: a D-SCOPE protocol. BMC Geriatr. 2018 Aug 27;18(1):194. doi: 10.1186/s12877-018-0875-3. PMID 30149798